CLINICAL TRIAL: NCT02701192
Title: Management of Coccydynia: A Prospective, Observational Study of Coccygectomy
Acronym: Coccyx
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 04-07-08B
Record Dates: First submitted 2016-02-11; First posted 2016-03-08 (Estimated); Results first posted 2021-06-14 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-06

CONDITIONS: Coccygodynia
Keywords: coccygodynia; coccygectomy; coccyx

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coccygectomy Treatment: Patients undergoing coccygectomy surgical procedure.
  Interventions: Other: Coccygectomy

INTERVENTIONS:
Other: Coccygectomy — Patient receiving coccygectomy surgery.

SUMMARY:
The purpose of the study is to analyze the outcomes of patients with coccygodynia (pain in and around the coccyx region) treated with coccygectomy (a procedure during which the coccyx is removed) and to report on the rate of complications of the procedure. The study will also aim to find pre-operative clinical predictors of good outcomes after coccygectomy. The investigators hypothesize that coccygectomy will not improve scores on the Short Form-36 (SF-36), Oswestry Disability Scale (ODI), tolerable sitting time, or Visual Analog Pain Scale (VAS). Also, the investigators hypothesize that there are no independent variables associated with improved outcomes.

DETAILED DESCRIPTION:
Coccygodynia can be a functionally limiting and painful disease with conservative treatment providing mixed results. When proper surgical indications are met, results seem to be promising. However, there is a lack of data in the literature to support surgical treatment. The case series reports currently in the literature are small and retrospective with ill-defined selection criteria. To date there has been no study prospectively following patients undergoing coccygectomy. This type of study could accurately obtain data prospectively. This information will help better guide the clinician through treatment of this disease.

All patients will be seen and enrolled through an outpatient spine specialty clinic of the senior author. Patients that meet the inclusion criteria will be offered enrollment in the study by a third party (clinical research assistant). Patients enrolled will then complete pre-treatment SF-36, Oswestry Disability Scale and a pain visual analog scale. Patients will be followed at 2 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years after treatment. Patients will complete the questionnaire containing the VAS and tolerable sitting time at all visits with SF-36 and Oswestry disability scale completed at one year post treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pain in the region of the coccyx
* Pain for greater than 2 months
* Tenderness to palpation over coccyx
* Radiographic abnormalities of the coccyx

  1. Hypermobility of greater than 25 degrees, posterior subluxation of a mobile segment, or a coccygeal spicule on sitting radiographs
  2. post-traumatic coccygodynia
* Failure of conservative treatment methods: 4 weeks of NSAIDS, seat cushion, and rest
* Partial coccygectomy

Exclusion Criteria:

* Coexisting low back pain
* Total previous coccyx surgery or previous lumbar fashion
* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will be seen and enrolled through an outpatient spine specialty clinic of Dr. Edward Hanley.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-09; Primary Completion 2015-12 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward N Hanley, MD, Principal Investigator — Carolinas Medical Center, Department of Orthopaedic Surgery
Locations (1):
- Carolinas Medical Center, Department of Orthopaedic Surgery, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 2007-2011, 98 patients underwent coccygectomy for chronic coccydynia. Included patients were over 18 years, had coccygeal pain and abnormality on physical and radiographic evaluation and had failed conservative management. Outcome measures were the Oswestry Disability Index (ODI), Visual Analog Scale (VAS) and the Short Form 36 (SF-36).
Period: Overall Study
Arm/Group | Coccygectomy Treatment
Started | 100
Completed | 94
Not Completed | 6
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Population: The study then evolved into a prospective observational case series of surgical treatment with total coccygectomy.
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 98
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.2 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 11
Etiology for Symptoms [Count of Participants; unit: Participants]
  Idiopathic | 47
  Trauma | 35
  Significant weight loss | 8
  Post-partum | 7
  Post floor surgery | 1
Co-morbidities [Count of Participants; unit: Participants]
  Pre-existing Spinal disorder | 17
  Non-spine related musculoskletal pathology | 37
  Psychiatric illness | 45
  Chronic pain | 28
  Genitourinary pain disorder | 3
  Other pain syndrome | 2
Coccydynia Pain Management [Count of Participants; unit: Participants]
  Prior Steroid Injection Therapy | 70
  Prior Opioid Use | 45

OUTCOME MEASURES:

1. Primary Outcome: Pain Change From Baseline at 2 Years
Description: Patients will complete the100mm Visual Analog Scale (VAS) at Baseline and 2 years after procedure. Patient will be instructed to indicate pain intensity by marking a 100mm line where one end, 0 indicates no pain and 100 indicates extreme pain on the other end.
Time Frame: Baseline,1 year and 2 years
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Pre-operative Baseline | 59.08 [54.06 to 64.1]
  One year | 19.35 [13.97 to 24.73]
  Two Years | 20.28 [14.64 to 25.92]

2. Primary Outcome: Patient Health Status- SF-36v2:Physical Functioning
Description: The SF-36 is on a 0-100 scale, with higher scores indicating a more favorable/better health state.
Time Frame: Baseline,1 year and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Baseline | 55.23 [48.65 to 61.81]
  One Year | 80.68 [74.67 to 86.99]
  Two Years | 79.24 [73.82 to 84.66]

3. Primary Outcome: Patient Health Status- SF-36v2: Role Functioning-Physical
Description: The SF-36 is on a 0-100 scale, with higher scores indicating a more favorable/better health state.
Time Frame: Baseline,1 year and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Baseline | 30.21 [22.07 to 38.35]
  One Year | 69.41 [59.98 to 78.84]
  Two Years | 70.12 [61.13 to 79.11]

4. Primary Outcome: Patient Health Status-SF-36v2: Role Functioning- Emotional
Description: The SF-36 is on a 0-100 scale, with higher scores indicating a more favorable/better health state.
Time Frame: Baseline,1 year and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Baseline | 54.17 [45.08 to 63.26]
  One Year | 86.99 [80.02 to 93.96]
  Two Years | 73.4 [64.67 to 82.13]

5. Primary Outcome: Patient Health Status-SF-36v2: Energy/Fatigue
Description: The SF-36 is on a 0-100 scale, with higher scores indicating a more favorable/better health state.
Time Frame: Baseline,1 year and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Baseline | 43.07 [38.21 to 47.93]
  One Year | 62.05 [56.86 to 67.24]
  Two Years | 60.78 [56 to 65.56]

6. Primary Outcome: Patient Health Status-SF-36v2: Emotional Well-being
Description: The SF-36 is on a 0-100 scale, with higher scores indicating a more favorable/better health state.
Time Frame: Baseline,1 year and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Baseline | 66.28 [62.02 to 70.54]
  One Year | 79.73 [75.81 to 83.65]
  Two Years | 77.44 [73.36 to 81.52]

7. Primary Outcome: Patient Health Status-SF-36v2: Social Functioning
Description: The SF-36 is on a 0-100 scale, with higher scores indicating a more favorable/better health state.
Time Frame: Baseline,1 year and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Baseline | 47.18 [42.11 to 52.25]
  One Year | 55.45 [51.26 to 59.64]
  Two Years | 55.81 [51.89 to 59.73]

8. Primary Outcome: Patient Health Status-SF-36v2: Pain
Description: The SF-36 is on a 0-100 scale, with higher scores indicating a more favorable/better health state.
Time Frame: Baseline,1 year and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Baseline | 39.95 [35.4 to 44.5]
  One Year | 70.34 [63.96 to 76.72]
  Two Years | 71.75 [66.06 to 77.44]

9. Primary Outcome: Patient Health Status-SF-36v2: General Health
Description: The SF-36 is on a 0-100 scale, with higher scores indicating a more favorable/better health state.
Time Frame: Baseline,1 year and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Baseline | 68.39 [64.4 to 72.38]
  One Year | 73.41 [68.61 to 78.21]
  Two Years | 69.31 [64.46 to 74.16]

10. Primary Outcome: Patient Health Status-SF-36v2: Health Change
Description: The SF-36 is on a 0-100 scale, with higher scores indicating a more favorable/better health state.
Time Frame: Baseline,1 year and 2 years
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Baseline | 45.31 [39.82 to 50.8]
  One Year | 81.4 [76.03 to 86.77]
  Two Years | 74.47 [68.98 to 79.96]

11. Primary Outcome: Lower Back Disability
Description: Oswestry Disability Index used to measure a patient's permanent functional disability. Scores range from 0 to 100. scores between 0 and 20 described as "minimal disability", scores between 21and 40 described as "moderate disability",scores between 41and 60 described as "severe disability",scores between 61 and 80 described as "crippled" and scores between 81 and 100 described as " bed bounded"
Time Frame: Baseline,1 year and 2 years
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
units on a scale
  Pre-operative Baseline | 39.07 [35.22 to 49.92]
  One Year | 15.39 [11.26 to 42.92]
  Two Years | 16.26 [12.59 to 19.93]

12. Secondary Outcome: Complication Rates
Description: Complication rates after coccygectomy surgery
Time Frame: Baseline,1 year and 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 94
Participants | 20

13. Secondary Outcome: Treatment Success
Description: Threshold for treatment success was based on a minimum clinically importance difference (MCID) of 20 points on the oswestry disability index at 2 year follow-up and an overall oswestry disability index score of <22 points.
Time Frame: Baseline,1 year and 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Coccygectomy Treatment
Number analyzed (Participants) | 98
Participants
  Treatment Success | 69
  Treatment Failure | 29

ADVERSE EVENTS:
Time Frame: Two years
Arm/Group | Coccygectomy Treatment
All-Cause Mortality (participants affected / at risk) | 0/98
Serious Adverse Events (participants affected / at risk) | 0/98
Other Adverse Events (participants affected / at risk) | 0/98

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-05-17): https://cdn.clinicaltrials.gov/large-docs/92/NCT02701192/Prot_SAP_000.pdf
  • Informed Consent Form (2011-05-10): https://cdn.clinicaltrials.gov/large-docs/92/NCT02701192/ICF_001.pdf